CLINICAL TRIAL: NCT01052506
Title: A Randomized, Blinded, Placebo-Controlled, Single Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of BIIB033 in Healthy Adult Volunteers
Brief Title: BIIB033 Single Ascending Dose Study in Healthy Volunteer Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 215HV101
Record Dates: First submitted 2010-01-15; First posted 2010-01-20 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Healthy
Keywords: Human volunteers
MeSH Terms: interventions — opicinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Single dose of saline solution (8 cohorts IV; 1 cohort SC)
  Interventions: Drug: Placebo
- BIIB033 (Experimental): Single, escalating doses of BIIB033 (8 cohorts IV; 1 cohort SC)
  Interventions: Drug: BIIB033

INTERVENTIONS:
Drug: BIIB033 — Single, escalating doses of BIIB033 (8 cohorts IV, 1 cohort SC)
  Other Names: Anti-LINGO-1 antibody
  Arms: BIIB033
Drug: Placebo — Single dose of placebo comparator (8 cohorts IV, 1 cohort SC)
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of single dose of BIIB033 administered to healthy adult volunteers.

DETAILED DESCRIPTION:
BIIB033 is an investigational product being developed to promote remyelination in subjects with multiple sclerosis (MS). This healthy volunteer study will evaluate safety and tolerability of a single dose of BIIB033.

ELIGIBILITY:
Inclusion Criteria:

* Must be in good health
* BMI of 18-30kg/m2
* Contraception required for at least 6 months after study drug administration

Exclusion Criteria:

* History of clinically significant disease or lab values
* Females of childbearing potentials
* Contraindication to brain MRI and/or lumbar puncture
* Treatment with any prescription medication within the 28 days prior to study entry
* Treatment with any over-the-counter products, including herbal and/or alternative health preparations and procedures within the 14 days prior to study entry
* Regular use of any tobacco product within 3 months prior to study entry

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2010-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Safety as measured by adverse event monitoring, laboratory assessments and MRI | up to 4 months
Tolerability as measured by adverse event monitoring, laboratory assessments and MRI | up to 4 months

SECONDARY OUTCOMES:
BIIB033 serum pharmacokinetics levels | up to 4 months
BIIB033 serum antibodies levels | up to 4 months
Exploratory blood, urine and CSF biomarkers | up to 4 months

CONTACTS AND LOCATIONS:
Locations (2):
- Research Site, Glendale, California, United States
- Research Site, Utrecht, Netherlands

REFERENCES:
- [Background] Tran JQ, Rana J, Barkhof F, Melamed I, Gevorkyan H, Wattjes MP, de Jong R, Brosofsky K, Ray S, Xu L, Zhao J, Parr E, Cadavid D. Randomized phase I trials of the safety/tolerability of anti-LINGO-1 monoclonal antibody BIIB033. Neurol Neuroimmunol Neuroinflamm. 2014 Aug 21;1(2):e18. doi: 10.1212/NXI.0000000000000018. eCollection 2014 Aug. PMID 25340070